CLINICAL TRIAL: NCT04083352
Title: The Effects of Exogenous Ketone Supplementation or a Ketogenic Diet in Individuals With PTSD
Brief Title: Ketone Supplementation in Individuals With PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 907405
Record Dates: First submitted 2019-08-05; First posted 2019-09-10 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-09

CONDITIONS: PTSD; Ketosis
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-week ketone supplementation (Experimental): Participants took a ketomax ketone salt supplementation for 6-weeks. They took 2 servings per day.
  Interventions: Dietary Supplement: Pruvit Ketomax Ketone Salt
- 6-week placebo supplement (Placebo Comparator): Participants took a placebo supplement for 6-weeks. The placebo was calorie, sodium, and flavor-matched to the experimental supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pruvit Ketomax Ketone Salt — 6-week supplementation with ketone salts
  Arms: 6-week ketone supplementation
Dietary Supplement: Placebo — Placebo was taken for 6-weeks and was calorie and flavor matched to the ketone salt supplement.
  Arms: 6-week placebo supplement

SUMMARY:
The purpose of this study is to determine if a 6-week period of ketone salt supplementation affects physiological, emotional, cognitive, and/or behavioral health markers in individuals with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PTSD

Exclusion Criteria:

* Pregnant, younger than 18 or older than 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Comprehensive Metabolic Panel | Pre- and Post- 6-week supplemental period
  Blood health marker
Change in Complete Blood Count | Pre- and Post- 6-week supplemental period
  Blood health marker
Change in Cognitive Performance | Pre- and Post- 6-week supplemental period
  ANAM test battery
Change in Blood Pressure | Pre- and Post- 6-week supplemental period
  Cardiovascular health measure
Change in Urinalysis | Pre- and Post- 6-week supplemental period
  Health measure

SECONDARY OUTCOMES:
Change in Insomnia | Pre- and Post- 6-week supplemental period
  Insomnia Severity Questionnaire
Change in Emotional Health | Pre- and Post- 6-week supplemental period
  Title: 12-Item Grit Scale; Construct: measures trait-level perserverance and passion for long-term goals; the scale for each question includes the following answers to check: Very much like me, mostly like me, somewhat like me, not much like me, not like me at all; Scoring: for questions 1, 4, 6, 9, 10, and 12 the following answers receive the associated number as a score: Very much like me (5), Mostly like me (4), Somewhat like me (3), Not much like me (2), Not like me at all (1). And questions 2, 3, 5, 7, 8, and 11 receive the following points for the checked answers: Very much like me (1 points), Mostly like me (2 points), Somewhat like me (3 points), Not much like me (4 points), Not like me at all (5 points). Add up all the points and divide by 12. The maximum score on this scale is 5 (extremely gritty) and the lowest score is 1 (not at all gritty).
Change in Emotional Health | Pre- and Post- 6-week supplemental period
  Title: Visual Analog Scales; Construct: measures the intensity or frequency of various symptoms; the scale is numerical with numbers from 0 to 10 lined horizontally and 0 indicates no symptom at all, 5 indicated neutral, and 10 indicates the highest feeling of the symptom. Symptoms asked included Hunger (0=not hungry at all, 10= very hungry), Satiety (0=don't feel full at all, 10=very full) , Mood (0= feel very down, 10= feel wonderful), Energy (0= very tired, 10=very energized), Focus (0= very distracted, 10=very focused), Alertness (0=non-coherent, 10= very aware of my surroundings)
Change in Emotional Health | Pre- and Post- 6-week supplemental period
  Mood Disorder Questionnaire
Change in alcohol use | Pre- and Post- 6-week supplemental period
  Alcohol Use Disorders Questionnaire
Change in PTSD | Pre- and Post- 6-week supplemental period
  PTSD Checklist for DSM-5
Change in PTSD | Pre- and Post- 6-week supplemental period
  Patient Health Questionnaire-9
Change in pain | Pre- and Post- 6-week supplemental period
  Pain Outcomes Questionnaire
Change in PTSD | Pre- and Post- 6-week supplemental period
  Adverse Childhood Experience Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided